CLINICAL TRIAL: NCT06338657
Title: A Window of Opportunity Study of Taxanes in Head and Neck Cancer
Brief Title: FID-007 Followed by Standard of Care Surgery in Head and Neck Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7H-23-5; NCI-2024-01367 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 7H-23-5 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2024-03-14; First posted 2024-03-29 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; Paclitaxel; Transurethral Resection of Bladder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (FID-007) (Experimental): Patients receive FID-007 IV over 30 minutes once a week for 3 weeks on days 1, 8, and 15 of a single 28 day cycle in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care surgery. Patients undergo CT or MRI during screening and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: PEOX-based Polymer Encapsulated Paclitaxel FID-007; Procedure: Tumor Resection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: PEOX-based Polymer Encapsulated Paclitaxel FID-007 — Given IV
  Other Names: FID 007; FID-007; FID007; Nanoencapsulated Paclitaxel FID-007; Paclitaxel in Polyethyloxazoline Polymer
Procedure: Tumor Resection — Undergo surgical resection

SUMMARY:
This phase I trial studies on how the PEOX-based polymer encapsulated paclitaxel FID-007 (FID-007) affects the immune cells around the tumor patients with head and neck squamous cell carcinoma. The active drug in FID-007 is paclitaxel, an established chemotherapy drug that has been shown to kill cancer cells. FID-007 is a packaged form of paclitaxel using a polyethylozaxoline (PEOX) polymer which may allow the drug to reach deeper into tumors and less into normal cells by being smaller. This study is being done to help identify future treatment options and better understand how to improve outcomes of patients with head and neck cancers after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To describe the phenotypical and functional changes of different T cell subsets within the tumor microenvironment after treatment with FID-007.

SECONDARY OBJECTIVES:

I. To describe the adverse events associated with neoadjuvant FID-007 prior to surgery for head and neck cancer.

II. To evaluate preliminary evidence of efficacy by describing the rate of major and complete pathologic response.

III. To describe the rates of locoregional recurrence and rate of distant metastasis at 2 years after surgery.

EXPLORATORY OBJECTIVE:

I. Explore association between pathologic response and phenotypical and functional changes in T cell subsets.

OUTLINE:

Patients receive FID-007 intravenously (IV) over 30 minutes once a week for 3 weeks on days 1, 8, and 15 of a single 28 day cycle in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care surgery. Patients undergo computed tomography (CT) or magnetic resonance imaging (MRI) during screening and blood sample collection throughout the study.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histopathologically / cytologically confirmed diagnosis of head and neck squamous cell carcinoma
* Sites of primary tumor allowed include the oral cavity and oropharynx only. Patients with recurrent disease that is amenable to surgery are eligible
* Patients may have any stage cancer amenable to surgical resection
* Patients must be able to provide an archival tissue specimen. Excisional biopsy or core needle biopsy specimens are allowed. Fine needle aspiration samples are not acceptable
* Patients with oropharynx cancer must have p16 negative disease
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Leukocytes ≥ 3,000/mcL
* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 100,000/mcl
* Hemoglobin ≥ 9 g/dl
* Total bilirubin ≤ 1.5 X institutional upper limit of normal
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/ Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 X institutional upper limit of normal
* Creatinine ≤ 1.5 X institutional upper limit of normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

  * A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy; or
    * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients with primary sites of the nasopharynx, salivary gland, or skin
* Patients that have been previously treated with taxane chemotherapies
* Patients that have previously received radiation to the site of planned surgery
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to FID-007 or other agents used in study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants
* Any diagnosis of immunodeficiency or patients receiving immunosuppressive therapy within 14 days of enrollment. Prednisone dose of ≤ 10mg is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the phenotypical and functional changes of different T cell subsets within the tumor microenvironment after treatment with FID-007 | Baseline up to 30 days
  Assessment of gene expression changes before and after the treatment with FID-007 by using paired biopsy samples by single cell-ribonucleic acid sequencing techniques. More specifically, the interested genes can be grouped as these four categories: (1) key immune checkpoint genes, including PD1, CTLA4, TIM3, LAG3, TIGIT, BTLA, VISTA, CD160, IDO, SIGLEC-15; (2) Gene signatures associated with T cell exhaustion: TOX, Blimp-1, Eomes, CD38, GZMB, GZMZ; (3) Gene signatures associated with T cell activation: CD3, CD28, NFAT, ZAP-70, CCR5, CCR7, and CXCR3, TCF-1; and (4) Gene signatures associated with T cell memory: CD45RO, CD62L, CCR7, IL-7R, BCL6, CD44, CXCR3.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Baseline up to 30 days
  A summary table at subject level focusing on grade 3 or higher treatment related AEs (as per Common Terminology Criteria for Adverse Events version 5.0) will be provided.
Major pathologic response rate | Up to 30 days
  Major pathologic response defined as 1-10% viable tumor on surgical specimen. Will be calculated based on the proportions that we calculated in the patient samples and their two-sided 95% confidence interval will also be estimated using Exact Clopper-Pearson method.
Complete pathologic response rate | Up to 30 days
  Complete pathologic response is defined as 0% viable tumor. Will be calculated based on the proportions that we calculated in the patient samples and their two-sided 95% confidence interval will also be estimated using Exact Clopper-Pearson method.
Rate of locoregional recurrence | Within 2 years of surgery (surgery will occur approximately 3-6 weeks after last dose of FID-007)
  Percentage of patients who develop local-regional recurrence (identification of disease growth) in the primary site or regional lymphatics based on imaging and/or clinical exam.
Rate of distant metastasis | Within 2 years of surgery (surgery will occur approximately 3-6 weeks after last dose of FID-007)
  The percentage of patients who develop distant metastasis within 2 years of surgery. Distant disease is cancer that is found in another part of the body that is far away from where the original (primary) tumor first formed.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Thomas, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California